CLINICAL TRIAL: NCT04192305
Title: Observational Study Evaluating the Impact of Lung Protective Ventilation (LPV) During Opioid Free Anesthesia (OFA) on Postoperative Oxygen Saturation.
Brief Title: Impact of LPV During OFA on Postoperative Oxygen Saturation.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, MD PhD, AZ Sint-Jan AV
Other Study IDs: OS impact LPV on SAT d OFA
Record Dates: First submitted 2019-12-02; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Oxygen Saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lung protective ventilation (LPV): lung protective ventilation low tidal volume, minimum PEEP and higher PEEP and lung recruitment based on total lung compliance, low inspiratory oxygen concentration and CPAP during extubation without prior suctioning inside the endotracheal tube.
  Interventions: Procedure: LPV
- routine lung ventilation (LV): ventilation and adapting PEEP, LRM and oxygen only when saturation drops.
  Interventions: Procedure: routine LV

INTERVENTIONS:
Procedure: LPV — LPV means tidal volume of 6 ml/kg, inspiratory-expiratory (I/E) ratio of 1/1, positive end expiratory pressure (PEEP) minimum 5 cmH20 and higher during laparoscopy in obese patients, Inspiratory oxygen concentration (FIO2) 40 % during maintenance and extubation while also giving CPAP. Lung recruitment maneuver (LRM) when lung compliance decreases below 40 ml/cmH2O.
  Groups: lung protective ventilation (LPV)
Procedure: routine LV — Give volume en frequency as required by end tidal carbon dioxide, PEEP and LRM only when saturation drops intra operative, no requirement to use low FIO2 and CPAP during extubation.
  Groups: routine lung ventilation (LV)

SUMMARY:
Observational study comparing patients with lung protective ventilation (LPV) following the consensus guidelines by Young C with patients getting routine lung ventilation, both during opioid free anesthesia (OFA).

DETAILED DESCRIPTION:
The paper by C Young et al describes the essential steps in protecting the lungs and preventing post operative pulmonary complications (PPC) like alveolar collapse.

Alveolar collapse can be measured by oxygen saturation drop when no oxygen therapy is given, when full neuromuscular block (NMB) reversal and no opioid is given intra and postoperative.

LPV means:

tidal volume of 6 ml/kg, inspiratory-expiratory (I/E) ratio of 1/1, positive end expiratory pressure (PEEP) minimum 5 cmH20 and higher during laparoscopy in obese patients, Inspiratory oxygen concentration (FIO2) max 80% during induction and max 40 % during maintenance and extubation. Extubation in an awake, full NMB reversed patient getting no opioids while giving continuous positive airway pressure (CPAP) during withdrawal of the tube. Lung recruitment maneuver (LRM) when lung compliance decreases below 40 milliliter per centimeter water. (ml/cmH2O)

ELIGIBILITY:
Inclusion Criteria:

* bariatric surgery
* morbid obesity ( BMI > 35)

Exclusion Criteria:

* patients with pre existing severe cardio-pulmonary diseases having oxygen saturation without oxygen below 94%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: bariatric surgery is performed in obese patients with BMI > 35
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
postoperative oxygen saturation | up to maximum 4 hours
  saturation is continuously measured in the post anesthetic area without giving oxygen until sat drops below 94%.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul Mulier, Principal Investigator — AZSint Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium